CLINICAL TRIAL: NCT02798718
Title: Effect of Whole Milk Intake on the Cardio-metabolic Risk Factors of Healthy Person With or Without Lactose Maldigestion
Brief Title: Whole Milk Intake and Cardio-metabolic Risk Factors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Liegang Liu, Professor, Huazhong University of Science and Technology
Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0214513214
Record Dates: First submitted 2016-05-24; First posted 2016-06-14 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Lactose Malabsorption; Cardiovascular Disease
MeSH Terms: conditions — Lactose Intolerance; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lactose digesters (Active Comparator): Participants in arm 1 are grouped as lactose digesters based on breath hydrogen test after a 25-g lactose load. The breath hydrogen excretion is less than 20 ppm.
  Interventions: Dietary Supplement: full-fat milk
- lactose maldigesters (Active Comparator): Participants in arm 2 are also grouped as lactose maldigesters based on breath hydrogen test after a 25-g lactose load. The breath hydrogen excretion is not less than 20 ppm.
  Interventions: Dietary Supplement: full-fat milk

INTERVENTIONS:
Dietary Supplement: full-fat milk — intake 250ml full-fat milk per day, do not intake any other dairy products

SUMMARY:
Milk is the source of high-quality protein, calcium, and other vitamins and minerals. Epidemiologic studies have linked high consumption of milk with risk of metabolic syndrome, T2DM, hypertension and obesity, which are independent risk factors of cardiovascular disease. However, milk contains disaccharide lactose, which may cause gastrointestinal problems in those adults with poor digestion. Recent studies have shown that subjects with intolerance to lactose tend to reduce their consumption of milk. Actually, consumption of 12g lactose (240ml milk) per day produces negligible symptoms in lactose intolerant. Furthermore, a dairy-rich diet could improve lactose intolerance because of colonic adaption to it. Lactose maldigestion would not be a restricting factor in milk intake. In general, the undigested lactose will be fermented by colonic bacteria into hydrogen, carbon dioxide, and short-chain fatty acids (SCFA: acetate, propionate, and butyrate). The SCFAs may have beneficial effects on human glucose and lipid metabolism, and the lactose fermentation may change the intestinal flora profile. But there are few studies evaluating effect of milk intake on health of people with lactose malabsorption or intolerance.This trial intend to study the effect of whole milk on cardio-metabolic risk factors of healthy person with or without lactose maldigestion.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 18 years of age
* Able to give informed connect

Exclusion Criteria:

* Unwilling to trial dietary intervention
* Pregnancy
* Known cardiovascular disease (stroke, ischemic heart disease and so on), diabetes, hypertension and any other chronic disease.
* Known gastrointestinal disease, such as Irritable Bowel Syndrome(IBS), functional bowel disease and so on.
* Evidence of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Changes in body weight | 4 weeks
Change in body composition (body fat mass and lean mass) | 4 weeks
  Body fat mass and lean mass measured by Bioelectric Impedance Analysis(BIA)
Changes in blood pressure | 4 weeks
  Systolic Blood Pressure and Diastolic Blood Pressure before and after milk intervention
Changes in blood lipids profile | 4 weeks
  Fasting plasma Total cholesterol, Low Density Lipoprotein, High Density Lipoprotein and triglycerides before and after milk intervention
Changes in fasting plasma glucose | 4 weeks
Changes in fasting plasma insulin | 4 weeks
Changes in fasting plasma C-peptide | 4 weeks
Changes in Homeostasis Model Assessment of Insulin Resistance(HOMA-IR) | 4 weeks
  Insulin sensitivity measure derived from fasting glucose and insulin

SECONDARY OUTCOMES:
Changes in pro-inflammatory markers | 4 weeks
  Fasting plasma C-reactive protein, interleukin-6 and tumor necrosis factor-α before and after milk intervention
Changes in markers of oxidative stress | 4 weeks
  Fasting plasma MDA, oxidized LDL before and after milk intervention
Biomarkers in urine | 4 weeks
Changes in fecal fat excretion | 4 weeks
Changes in fecal short chain fatty acids (SCFA) | 4 weeks
  Fecal acetate, propionate, butyrate before and after milk intervention

CONTACTS AND LOCATIONS:
Overall Officials: Liegang Liu, PhD, Study Chair — Huazhong University of Science and Technology
Locations (1):
- Huazhong University of Science and Technology, Wuhan, Hubei, China